CLINICAL TRIAL: NCT05439733
Title: Planned Mode of Delivery After Caesarean: a Comparative Prospective National Population-based Cohort Study
Acronym: CICAMODA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-A00514-39
Record Dates: First submitted 2022-06-02; First posted 2022-06-30 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Scarred Uterus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Exposed group: Women with a history of cesarean section and with a base-line attempt after planned cesarean section (TVBAC).
  Interventions: Other: Questionnaire completion
- Non-exposed group: Women with a history of cesarean section and scheduled cesarean section after cesarean section (CPAC).
  Interventions: Other: Questionnaire completion

INTERVENTIONS:
Other: Questionnaire completion — Women will be asked to complete questionnaires 6 weeks after delivery

SUMMARY:
In women with one previous caesarean, the choice of mode of delivery is determined by a shared decision-making process between the women and the obstetrician, with the two options being a trial of labour after caesarean (TOLAC) or an elective repeat caesarean delivery (ERCD).

To date, the scientific literature has reported of higher perinatal morbidity-mortality with TOLAC, although with low absolute risks and discordant results about maternal morbidity-mortality. These studies suffer from limitations, as they include women with more than one previous caesarean or with high rates of failed TOLAC, which are two risk factors for uterine rupture, and the definition of planned versus effective mode of delivery is not precise in most studies.

However, scientific societies recommend that most women with one previous caesarean should be offered TOLAC because of the low absolute perinatal risk of this option and the high maternal and perinatal risk associated with an ERCD in the short- and long-term.

Conversely, the investigators hypothesise that TOLAC would be not inferior to ERCD in women with one previous caesarean in terms of perinatal morbidity-mortality.

DETAILED DESCRIPTION:
Primary and secondary objectives :

The primary objective is to evaluate the non-inferiority of TOLAC compared to ERCD on the perinatal morbidity-mortality rate. The secondary objectives are to compare between the TOLAC and ECRD groups: the maternal morbidity-mortality rate, care trajectories of women and child one year after delivery, the uterine rupture rate, pain experienced during delivery, the breastfeeding rates at the time of hospital discharge and at 6-weeks postpartum, the satisfaction, the quality of life, and the bonding of women at 6-weeks postpartum, the risk of postnatal depression, and the post-traumatic stress disorder at 6-weeks postpartum, the medical resource costs and perform a cost-effectiveness analysis or a cost-minimization analysis depending on the result on the primary endpoint, the risk perception of women and of the obstetrician about the course of delivery: at the time of the shared decision-making process with the obstetrician of their planned mode of delivery, two days after delivery, and at 6-weeks postpartum (ancillary study CICAMODA Risk), and the risk of urinary incontinence at 12 months postpartum (ancillary study CICAMODA PP).

Methods :

* Design : the investigators plan a national multicentre prospective observational cohort study.
* General procedure : after admission of the women in the labour ward and within the 72 hours after birth, obstetricians will inform women about the study and determine whether or not they object to participate, in accordance with French law. The investigators will collect data about characteristics of the women, the previous caesarean delivery, the planned mode of delivery, the pregnancy, the course of labour, and postpartum data.
* Schedule : the investigators plan a 12-month inclusion period to obtain a complete view of French practices in planned mode of delivery after one previous caesarean delivery thanks to this observational study. The duration of the follow-up period will be 12-months for each included woman.
* Sample size : thanks to data of 2016 National Perinatal Survey, the investigators assume that TOLAC will be planned in 68.9% of French women with one previous caesarean and ERCD in the remaining 31.1%.

From an analysis of the literature, the investigators estimate that the perinatal morbidity-mortality rate is 0.9% in the ERCD group. The noninferiority boundary based on clinical evidence and an expert committee has validated an estimated rate of perinatal morbidity-mortality of 1.4% in the TOLAC group. According to these assumptions and with a power of 80% and a one-sided alpha risk of 2.5%, the number of women to be included is 4343 in the ERCD group and 9669 in the TOLAC group, i.e. a total of 14,012 women. With anticipation that 5% of women will provide incomplete data to define the primary outcome, 14750 women will be needed.

During the inclusion period, the investigators except to include 16800 women, which will provide enough power to investigate the non-inferiority of TOLAC in terms of perinatal morbidity-mortality.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women age of 18 years or older
* Women admitted to the labour ward at gestational age ≥ 34 weeks
* Women with a singleton pregnancy
* Women with one previous caesarean delivery
* Computer savvy-women Exclusion Criteria:

Exclusion criteria :

* Women who oppose to participation in the study
* Age < 18 years
* Women admitted to the labour ward at gestational age < 34 weeks
* Women with multiple pregnancy
* Women with more than one previous caesarean or more than one uterine scar
* Women who do not understand the French language
* Women under judicial protection

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant women age of 18 years or older
Study Population: Pregnant women age of 18 years or older
Sampling Method: Non-Probability Sample
Enrollment: 16800 (Estimated)
Dates: Start 2022-08-02 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint will be the perinatal morbidity-mortality rate | From admission and maximum 28 days after delivery
  Composite measure of:
  * Perinatal death (any foetal death or death of a liveborn infant before hospital discharge [excluding lethal congenital anomalies])
  * Birth trauma
  * SARNAT Stage 2 or 3 hypoxic ischemic encephalopathy
  * Perinatal asphyxia, which is fulfilment of at least one of the following criteria:
    * Severe biological signs: Arterial or venous cord blood pH < 7,0 or Base deficit ≥ 16 mmol/L or Lactate ≥ 11 mmol/L
    * Or 7.0 < pH ≤ 7.15, or 10 ≤ base deficit < 16 mmol/L, ou 8 ≤ lactates < 11 mmol/l, or not available but with:
    * Perinatal event (severe non reassuring fetal hearth rate, cord prolapse, uterine rupture, maternal trauma or cardio-respiratory arrest
    * Or sudden change of fetal hearth rate
    * Or 10 minutes Apgar score of 5 or less or assisted ventilation initiated at birth and continued for at least 10 minutes
    * Admission to intensive care with intratracheal intubation or need for ventilation
  * Length of stay in Neonatal Intensive

SECONDARY OUTCOMES:
Maternal morbidity-mortality rate | From admissionand maximum 15 days after delivery
  Maternal death
  * Severe postpartum haemorrhage (blood loss ≥ 1000 mL)
  * Blood transfusion
  * Obstetrical anal sphincter injury (stages 3 or 4 of the Royal College of Obstetricians and Gynaecologists classification of perineal tears)
  * Intensive care unit admission
  * Damage to the bladder, ureter or bowel requiring repair
  * Wound infection or wound dehiscence (requiring prolongation of hospital stay)
  * Readmission to the operating room
  * Hysterectomy
  * Deep vein thrombosis, thrombophlebitis, or pulmonary embolus requiring anticoagulant therapy
  * Proven endometritis (positive vaginal bacteriology) or proven postpartum sepsis (positive blood cultures)
  * Prolongation of hospital stay > 15 days
Uterine rupture rate | During the surgery and confirmed by an adjudication committee.
  Defined as a clinically significant rupture involving the full thickness of the uterine wall and requiring surgical repair
Breastfeeding rate at the time of hospital discharge | Between day 3 and day 5
  Breastfeeeding rate
Felt pain during delivery | 6-weeks postpartum
  The felt pain during delivery will be evaluated thanks to numeric scale (0 to 10) and how was dealt the pain by the team of care. A low score means that the patient's postpartum pain is low. On the contrary, the higher the score, the greater the pain.
Breastfeeding rate | 6-weeks postpartum
  The breastfeeding will be evaluated by the following questions:
  Do you breastfeed your baby at the present time? Do you give bottles to your baby at the present time? The maternal satisfaction will be evaluated as previously reported in this specific clinical situation.
Evaluate the satisfaction | 6-weeks postpartum
  Thanks to Likert scales, we will evaluate the satisfaction about the previous caesarean delivery, about the most recent delivery, about the recovery after the previous caesarean delivery and after the most recent delivery, and about the most recent delivery in comparison with the previous caesarean delivery.
Evaluate the quality of life | 6-weeks postpartum
  The quality of life will be evaluated thanks to the Short-Form 12 (SF-12) as recommended. The choice of the 12 items version is justified by the feasibility (acceptability by the postpartum women).
  A low score means that the patient's quality of life is low. The higher the score, the higher the quality of life.
Risk of postnatal depression, and post-traumatic stress disorder | 6-weeks postpartum
  (French version Edinburgh Postpartum Depression Scale EPDS)81. The score per question varies from 0 to 3. The higher the score, the greater the risk of postnatal depression and post-traumatic stress disorder.

CONTACTS AND LOCATIONS:
Overall Officials: François CREMIEUX, Study Director — ASSITANCE PUBLIQUE HOPITAUX MARSEILLE; Julie BLANC, Principal Investigator — ASSITANCE PUBLIQUE HOPITAUX MARSEILLE
Locations (1):
- Assistance Publique Hôpitaux Marseille, Marseille, Bouches-du-rhône, France